CLINICAL TRIAL: NCT07141303
Title: Intra-arterial Methylprednisolone After Successful Endovascular Thrombectomy Anterior Circulation Large Vessel Occlusion
Acronym: IMPACT-LVO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Collaborators: The First people's hospital of Xian Yang (Unknown); First People's Hospital Of Tianshui (Unknown); XD Group Hospital (Unknown); Xi'an Aerospace General Hospital (Unknown); First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K202508-15
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The methylprednisolone sodium succinate group (Experimental): The methylprednisolone sodium succinate group patients will receive intra-arterial methylprednisolone sodium succinate 40mg immediately after the recanalization. Then, intravenous administration with methylprednisolone sodium succinate 2mg/kg in the next 3 days.
  Interventions: Drug: The methylprednisolone sodium succinate
- The placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: The methylprednisolone sodium succinate — Patients will receive intra-arterial methylprednisolone sodium succinate 40mg immediately after the recanalization from thrombectomy in anterior circulation large vessel occlusion. Then, intravenous administration with methylprednisolone sodium succinate 2mg/kg in the next 3 days.
  Arms: The methylprednisolone sodium succinate group
Drug: Placebo — The placebo group patients will receive intra-arterial and intravenous sterile water for injection.
  Arms: The placebo group

SUMMARY:
The purpose of IMPACT-LVO trial is to investigate the efficacy and safety of early adjunctive intra-arterial combined with intravenous administration methylprednisolone sodium succinate after successful endovascular thrombectomy in anterior circulation large vessel occlusion patients.

This is a multicenter, randomized, double-blind, placebo-controlled trial. Acute ischemia stroke patients with anterior circulation large vessel occlusion within 24 hours from last known well will be screened for this trial. Successful recanalization after mechanical thrombectomy (eTICI 2b-3) patients will be randomized 1:1 to either methylprednisolone sodium succinate group or placebo group. The methylprednisolone sodium succinate group patients will receive intra-arterial methylprednisolone sodium succinate 40mg immediately after the recanalization. Then, intravenous administration with methylprednisolone sodium succinate 2mg/kg in the next 3 days. The placebo group patients will receive intra-arterial and intravenous sterile water for injection.

The shift on modified Rankin Scale score is designed to detect in the present trial. A sample size of n = 1010 patients (n=505 per group) is required. The intention-to-treat principle will be applied to the primary analysis, therefore, to safeguard against dilution of the treatment effect associated with an approximate 5% non-adherence rate (due to loss to follow-up, consent withdrawal and other reasons), we planned to enrol n=1060 patients (n=530 per group) for this study. The findings of IMPACT-LVO are likely to have a direct impact on clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old; 2) The time from onset to randomization was within 24 hours; 3) Large vessel occlusive stroke in the anterior circulation confirmed by CTA/MRA/DSA (Including intracranial segment of internal carotid artery, M1 or M2 segment of middle cerebral artery) and the vessel responsible for the signs and symptoms of acute ischemic stroke; 4) NIHSS score >= 6 points 5) Alberta Stroke Program Early Diagnosis (ASPECTS) score of NCCT >=3; 6) Successful endovascular thrombectomy (eTICI 2b50-3) 7) Written informed consent signed by patients or their family members

Exclusion Criteria:

1. Intracranial hemorrhage confirmed by computed tomography (CT) or magnetic resonance imaging (MRI);
2. Prestroke mRS score >= 2
3. pregnant or lactating patients
4. Allergy to iodinated contrast media, or methylprednisolone sodium succinate
5. Participating in other clinical research;
6. Inherited/acquired hemorrhagic diathesis (coagulation factor deficiency) or oral anticoagulation with international normalized ratio (INR) >1.7
7. History of major bleeding within the past 1 month (gastrointestinal/genitourinary hemorrhage)
8. Chronic hemodialysis and severe renal insufficiency (glomerular filtration rate < 30ml/min/1.73m^2 or serum creatinine > 220μmol/L (2.5mg/dl));
9. Terminal illness with life expectancy <6 months;
10. Blood glucose < 2.8mmol/L (50mg/dl) or > 22.2mmol/L (400mg/dl);
11. Intracranial aneurysm, arteriovenous malformation, or space-occupying brain tumor with mass effect on imaging
12. Active systemic infectious disease
13. Anticipated inability to complete follow-up
14. Intraoperative DSA showed vascular perforation, dissection, and contrast extravasation;
15. Puncture to recanalization was more than 90 minutes; Total thrombectomy passes >3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Shift in the distribution of mRS scores | 90 days
Incidence of symptomatic intracranial hemorrhage | 48 hours
Mortality | 90 days

SECONDARY OUTCOMES:
The proportion of mRS score 0 to 4 | 90 days
The proportion of mRS score 0 to 3 | 90 days
The proportion of mRS score 0 to 2 | 90 days
mRS scores | 1 year
The incidence of malignant brain edema | within 48 hours
Changes of NIHSS score | 5-7 days after surgery
EQ-5D scale score | 90 days
EQ-5D scale score | 1 year
Proportion of patients with any radiologic intracranial haemorrhage | within 48 hours after treatment
Proportion of patients with pneumonia | within 7 days after the treatment
Proportion of patients with gastrointestinal haemorrhage | within 7 days after treatment
Incidence of non-hemorrhagic serious adverse events | within 7 days after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Related papers published five years later, the IPD will be shared on ResMan.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Related papers published five years later, the IPD will be shared on ResMan.